CLINICAL TRIAL: NCT04280770
Title: Surgical Techniques for Epiretinal Membrane Removal in Pars Plana Vitrectomy: A Comparative Study Between 20-Gauge and 23-Gauge Vitrectomy
Brief Title: 23-gauge Pars Plana Vitrectomy With Silicone Oil Injectionsilicone Oil Injection With Surgical
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, khaled hamdi elbaklish, Clinical Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FWA000017585 FMASU 25/2017
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Retinal Detachment
Keywords: retina; silicone; laser; break; vitrectomy
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Intervention Model Description: Fifty participants were assigned and divided into two groups. Participants without RD after SO removal was recruited into group A-NRD, and participants with RD after SO removal was recruited into group B-RD.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Each of the recruited patients were assigned a study number and randomized in accordance with a simple block randomization scheme.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non retinal detachment group (Sham Comparator): 35 participants did 23 vitrectomy followed for 3-6 months. After that, we removed the oil and followed them for 6 weeks.
  Interventions: Procedure: 23 PARS PLANA VITRECTOMY
- retinal detachment group (Active Comparator): 15 participants did 23 vitrectomy followed for 3-6 months. After that, we removed the oil and followed them for 6 weeks.
  Interventions: Procedure: 23 PARS PLANA VITRECTOMY

INTERVENTIONS:
Procedure: 23 PARS PLANA VITRECTOMY — We performed a three-port vitrectomy: one infusion trocar and two instruments trocars. Non-contact wide-angle viewing systems (Resight- Biom) have a viewing field of 60-130° was used. Put 23 needle attached to the automated pump for silicone oil extraction. Strict examination of the retina to detect new breaks or untreated breaks. Closure of the sclerotomies.
  Other Names: SILICONE OIL REMOVAL

SUMMARY:
Objective: to evaluate anatomical and visual outcomes of 23-gauge vitrectomy for retinal detachment with silicone oil injection in fifty cases. The rate of recurrence, the incidence of proliferative vitreoretinopathy (PVR) and the value of risk factors.

Participants and Methods: fifty cases with RD with mixture of epiretinal and subretinal membranes were collected. Pars plan vitrectomy, 23gauge vitrectomy were done to these cases, then silicone oil removed 6 weeks after primary surgery.

Main Outcome Measures: The anatomical success rate,the failure rate ,the rate of retinal breaks in both groups, and reproliferation rate.

DETAILED DESCRIPTION:
50 Patients were included if they had retinal detachment, moderate degrees of PVR, PVR ≥ Grade C, previous buckle surgery and pseudophakia. A good and correct assessment of the detached retina was done. Investigator followed the Lincoff rules to find the retinal breaks. Investigator performed a three-port vitrectomy: one infusion trocar and two instruments trocars. Non-contact wide-angle viewing systems (Resight- Biom) have a viewing field of 60-130° was used. Investigator used Perfluorocarbon liquid (PFCL) for attaching the retina with its gravity. Then performing PFCL against air exchange.The retina will be attached under air tamponade. Laser photocoagulation was performed in the air-filled eye.

Investigator applied the laser effects confluently surrounding all retinal breaks. Then silicone oil (1000 centistokes) was injected as a final step and permanent tamponade.After 3-6 months investigator removed the silicone and examined the retina for 6 weeks after surgery to detect the recurrent cases.

ELIGIBILITY:
Inclusion Criteria:

* they had retinal detachment,
* moderate degrees of PVR
* PVR ≥ Grade C
* previous buckle surgery
* pseudophakia.

Exclusion Criteria:

* the retinal tear was greater than 90 degrees
* presence of intravitreal foreign body
* previous vitrectomy done before
* if follow-up data were unavailable for a minimum follow-up of 6 months following the final retinal procedure.

Ages: 23 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-01-30 (Actual); Primary Completion 2013-03-11 (Actual); Study Completion 2013-03-30 (Actual)

PRIMARY OUTCOMES:
success rate | 42 days
  success rate after first RD surgery and silicone oil removal
The failure rate | 42 days
  The failure rate after silicone oil removal
number of surgical interference | 4 years
  numbers of vitrectomies done after silicone oil removal

SECONDARY OUTCOMES:
lower retinal breaks | 4 years
  The rate of lower retinal breaks in RD group versus the rate of lower retinal breaks in NRD group was

IPD SHARING:
Plan to Share IPD: No
no plan till now